CLINICAL TRIAL: NCT00004056
Title: Treatment of Newly Diagnosed Childhood AML Using a Timed-Sequential Remission Induction and Consolidation Followed by Single Dose Melphalan With Peripheral Stem Cell Rescue: A POG Pilot Study
Brief Title: Combination Chemotherapy Followed by Melphalan and Peripheral Stem Cell Transplantation in Treating Children With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9822; POG-9822; CDR0000067253
Record Dates: First submitted 1999-12-10; First posted 2004-05-20 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia
Keywords: untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood acute monoblastic leukemia and acute monocytic leukemia (M5); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myelomonocytic leukemia (M4); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); childhood acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Monocytic, Acute | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Asparaginase; Cytarabine; Daunorubicin; Melphalan; Thioguanine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemo + STEM cell (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Drug: asparaginase; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: melphalan; Drug: thioguanine; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; GCSF; Neupogen®; NSC #614629
Drug: asparaginase
  Other Names: E. coli; Elspar; NSC #109229
Drug: cytarabine
  Other Names: cytosine arabinoside; AraC; Cytosar; NSC #063878
Drug: daunorubicin hydrochloride
  Other Names: daunomycin; DNR; Cerubidine; NSC #82151
Drug: melphalan
  Other Names: L-phenylalanine mustard; L-PAM; L-sarcolysin; Alkeran; NSC #008806
Drug: thioguanine
  Other Names: 6-thioguanine; 6-TG; NSC #000752
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy followed by melphalan and peripheral stem cell transplantation in treating children who have newly diagnosed acute myeloid leukemia that has not been treated previously.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility and toxicity of timed sequential remission induction and consolidation in children with newly diagnosed acute myeloid leukemia. II. Determine the feasibility and toxicity of a single high dose of melphalan with peripheral blood stem cell rescue following an intense timed sequential induction and consolidation in these children.

OUTLINE: This is a multicenter study. Remission induction: Patients receive daunorubicin IV over 15 minutes on days 1-3, cytarabine IV continuously on days 1-7, oral thioguanine daily on days 1-7, and cytarabine intrathecally (IT) on day 1. Cytarabine IV over 3 hours is administered every 12 hours on days 10-12. Filgrastim (G-CSF) is administered IV or subcutaneously (SQ) beginning on day 13 and continuing until blood counts recover. On approximately day 28, patients undergo a bone marrow aspirate and biopsy to assess response. Patients who have attained an M1 or M2a status proceed to consolidation or, if a 5/5 or 6/6 HLA matched sibling donor is available, proceed to allogeneic bone marrow transplantation. Patients with greater than 25% blasts go off study. Consolidation 1: Patients receive daunorubicin IV over 15 minutes on days 1 and 2, cytarabine IV over 3 hours every 12 hours on days 1, 2, 8, and 9, and asparaginase on days 2 and 9. G-CSF IV or SQ begins on day 10 and continues until blood counts recover. Consolidation 2: Patients receive cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5. G-CSF IV or SQ begins on day 6 and continues until blood counts recover. Peripheral blood stem cells (PBSC) are collected after the second course of consolidation. Consolidation 3: Treatment is repeated as in consolidation 1. Patients who remain in morphologic remission after consolidation 3 proceed with therapy. Patients receive melphalan IV over 30 minutes on day -2, then PBSC are reinfused on day 0. G-CSF IV or SQ begins on day 1 and continues until blood counts recover. Patients are followed every 6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, previously untreated primary acute myeloid leukemia (AML) Isolated granulocytic sarcoma (myeloblastoma) allowed Patients with cytopenias and bone marrow blasts greater than 5% but less than 30% eligible only if there is karyotypic abnormality characteristic of de novo AML (t(8;21), inv16, t(9;11), etc.) OR unequivocal presence of megakaryoblasts No acute promyelocytic leukemia (M3) No Down syndrome

PATIENT CHARACTERISTICS: Age: 21 and under Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Uric acid no greater than 8.0 mg/dL Cardiovascular: Cardiac function normal by echocardiogram Pulmonary: No uncontrolled, life threatening pneumonia Other: No uncontrolled, life threatening sepsis or meningitis Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: No prior therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 1999-10; Primary Completion 2002-10 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Feasibility and toxicity of an intensive regimen that uses timed-sequential therapy | Length of study
  To determine the feasibility and toxicity of an intensive regimen that uses timed-sequential therapy as a strategy for both remission induction and consolidation of newly diagnosed children with AML.
Feasibility and toxicity of a single high dose of melphalan with peripheral stem cell rescue | Length of study
  To test the feasibility and toxicity of a single high dose of melphalan with peripheral stem cell rescue following an intense timed-sequential induction and consolidation.

SECONDARY OUTCOMES:
Make observations regarding PCR evidence of Minimal Residual Disease | Length of study
  To make observations regarding PCR evidence of Minimal Residual Disease in patients with relevant specific translocations who obtain a clinical remission.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Hurwitz, MD, Study Chair — Maine Children's Cancer Program at Barbara Bush Children's Hospital
Locations (20):
- United States (19):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Children's Hospital and Health Center, San Diego, California
  - Nemours Children's Clinic, Jacksonville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Tomorrows Children's Institute, Hackensack, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Montreal Children's Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Result] Hurwitz CA, Chang M, Graham M, et al.: Timed-sequential remission induction and intensification followed by stem cell rescue for childhood AML -a POG pilot study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1553, 2002.